CLINICAL TRIAL: NCT04938102
Title: Role of EndoFLIP in the Diagnostic Paradigm of Esophagogastric Junction Outflow Obstruction
Acronym: EndoFLIP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative-not IRB approved
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Reza Hejazi, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY00147450
Record Dates: First submitted 2021-06-21; First posted 2021-06-24 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Esophagogastric Junction Disorder
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Abnormal DI - Control (No Intervention): Patients' whose distensibility index is measured <2.8 will receive no intervention.
- Abnormal DI - Botox (Active Comparator): Patients' whose distensibility index is measured <2.8 will be injected with 100 units of botulinum toxin in the lower esophageal sphincter (25 units in each quadrant).
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]
- Normal DI - Control (No Intervention): Patients' whose distensibility index is measured >2.8 will receive no intervention.

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Botox] — Injection of 100 units of botulinum toxin into the lower esophageal sphincter (25 units in each quadrant).
  Arms: Abnormal DI - Botox

SUMMARY:
The aim of this project is to identify if EndoFLIP can categorize and change the diagnosis in patients with EGJOO and if categorization with EndoFLIP can predict the response to treatment with botulinum toxin at 12 weeks post procedure. Our hypothesis is that there will be greater symptom resolution in the treatment versus control in the abnormal DI category. In addition, we hypothesize there will be less symptom resolution in the control group with an abnormal DI as compared to those with a normal DI who also receive no treatment.

DETAILED DESCRIPTION:
Esophagogastric Outflow Obstruction (EGJOO) is a newer diagnosis in which some patients' symptoms resolve spontaneously or with conservative treatment, while others require treatment with botulinum toxin injected into the lower esophageal sphincter. Currently, there is no way to distinguish these two groups of patients upon diagnosis. EndoFLIP (endolumenal functional lumen imaging probe) is a new technology that can measure the distensibility index (DI) of the lower esophageal sphincter. Data has suggested that normal and abnormal DI measurements can categorize these patients and guide treatment course (1). Our study looks to confirm this finding.

1. Elsbernd et al. Clinical characteristics and treatment response of esophagogastric junction outflow obstruction. Gastroenterology 2019;156(6):S-1017.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with esophagogastric junction outflow obstruction by high resolution manometry

Exclusion Criteria:

* previous upper gastrointestinal surgery
* significant medical co-morbidities
* eosinophilic esophagitis
* severe reflux esophagitis (LA-classification C or D)
* large hiatal hernia
* patients experiencing significant weight loss suspicious for malignancy
* Vulnerable populations such as cognitively or decisionally impaired individuals, children, pregnant women, prisoners, and students or employees of the University of Kansas Health System or Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Symptom Resolution | 12 weeks.
  The primary endpoint is the proportion of patients with complete symptom resolution at 12 weeks (Eckardt score < 3) post procedure in each group.

SECONDARY OUTCOMES:
Percent change in symptom score | 12 weeks.
  The secondary endpoint is the percent change in symptom score at 12 weeks in each group.
Mean symptom scores | 12 weeks.
  The secondary endpoint is the change in mean symptom score in each group at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Hejazi, MD, Principal Investigator — University of Kansas Medical Center

IPD SHARING:
Plan to Share IPD: No